CLINICAL TRIAL: NCT06035666
Title: REducing Stress and Improving professionaLs' vItality Using innovativE iNtervenTions
Acronym: RESILIENT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Erasmus Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Principal Investigator, dr. Laura C. G. de Graaff-Herder, Principal Investigator, Erasmus Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 9642
Record Dates: First submitted 2023-09-04; First posted 2023-09-13 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Mental Health Issue; Healthy Lifestyle; Stress, Psychological
Keywords: eHealth; Vitality; Stress; Heath care workers; App; Your World
MeSH Terms: conditions — Stress, Psychological; Alzheimer Disease

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial
Masking Description: Not possible
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Sham Comparator): Control app
  Interventions: Other: Control app
- Intervention (Experimental): Your World (vitality session + app)
  Interventions: Other: Your World

INTERVENTIONS:
Other: Your World — Your World consists of a vitality session and use of the Your World app
  Arms: Intervention
Other: Control app — Control app, no effect on stress/vitality
  Arms: Control

SUMMARY:
Introduction Up to half of hospital employees worldwide are experiencing symptoms of burnout. Therefore, interventions to improve mental health among hospital workers are urgently needed. Your World is an inexpensive and easy-to-use intervention that aims to reduce stress and increase resilience among hospital employees. Your world uses a blended approach, which includes a real-life personal session and challenges in the Your World app (for smartphone).

Hypothesis The investigators hypothesize that Your World will improve resilience and well-being and reduce stress among hospital employees.

Research objectives Main objective

- Does Your World reduce stress among hospital employees as measured by the PSS-10?

Design Randomised controlled trial

Population Employees of the Erasmus University Medical Center including students and volunteers

Methods and study procedures Five hundred participants will be randomized 1:1 to receive either Your World (intervention) or the control app (control). In the intervention group, subjects will participate in one 'vitality session' before installing the app. At baseline and after 3 months hair samples questionnaires will be collected among the participants of both groups. At 6 months, same questionnaires will be collected.

Burden and risks There are no risks associated with participation in this study. The questionnaires can be filled out online in 15 minutes, hair collection takes 5 minutes. The vitality sessions take 1 hour and the use of the app takes 5 minutes a day.

DETAILED DESCRIPTION:
1. Introduction and rationale Hospital employees are under a lot of pressure due to a large physical and emotional workload and time constraints (1). This may lead to exhaustion, psychological or physical distress and eventually burnout. Maslach et al. (2) have defined three dimensions of burnout: exhaustion, cynicism/depersonalization and sense of inefficacy/low personal accomplishment. Burnout among health care professionals has been an under-recognized and under-reported problem. There is increasing data about burnout and mental vitality among health care workers; up to half of hospital employees are experiencing symptoms of burnout (3-7). Psychological problems among health care workers can cause decreased job satisfaction, decreased efficiency and productivity, absenteeism, abandonment of the medical profession and even poor quality of care and impaired patient safety (4,8-11). Several interventions have been developed to promote well-being and reduce psychological problems among health care workers, including coaching programs and mindfulness and cognitive-behavioral therapy-based interventions (12,13). Although effective, these programs are usually expensive and time-consuming.

   To increase availability (and to reduce costs) of mental support for healthcare professionals, Your World has been developed. Your World is designed to improve employees' well-being and resilience by implementing new habits according to the 'Healthy Mind Platter' (HMP) (14). Contrary to most existing interventions, Your World is inexpensive and time-efficient, taking only a couple of minutes a day. The healthy mind platter consists of seven neuro-cognitive activities or 'ingredients' that are important for stress reduction: physical time (exercise), sleep time, focus time (planning moments for work or hobbies without interruptions), time in (self-reflection), down time (moments without scheduled tasks), play time (playing and humor) and connecting time (social interaction or time spent with nature). In the Your World app, an eighth dimension was added: earth time, which is related to nature connectedness and pro-environmental behavior.

   Through weekly challenges (trying out a new habit) and encouraging messages, the app motivates the users to implement new HMP activities into their daily life, in order to improve mental well-being.

   The investigators hypothesize that Your World will improve resilience and mental vitality and reduce stress among health care employees. Eventually, this will reduce negative psychological outcomes like burnout and its practical consequences (absenteeism, dropout).
2. Objective(s)

   Main objective

   - Does Your World reduce stress among hospital employees as measured by the PSS-10?

   Secondary objectives
   * Does Your World reduce stress among hospital employees as measured by hair cortisol levels?
   * Does Your World improve vitality among hospital employees as measured by the Vita-16?
   * Which factors (e.g. age, gender, job and department) influence stress and vitality of hospital employees?
   * What is the relation between different measurements (i.e. PSS-10, vita-16, vitality scores, mood scores and hair cortisol) of stress and vitality?
   * Which factors (e.g. stress, vitality, age, gender, job) influence the use of the Your World app?
3. Study type

   3.1 Study type:

   Prospective randomized controlled trial
4. Methods

4.1 Methods In total, 500 participants will be randomized to the intervention or the control group. Participants in the intervention group will undergo a vitality session and receive a code needed to download and use the Your World app. The control group will not participate in vitality sessions, but they will receive access to the control app. In both groups, hair samples and stress / vitality questionnaires will be collected at baseline and after 3 months. Questionnaires will be collected again after 6 months.

References

1. Dubale BW, Friedman LE, Chemali Z, Denninger JW, Mehta DH, Alem A, Fricchione GL, Dossett ML, Gelaye B. Systematic review of burnout among healthcare providers in sub-Saharan Africa. BMC Public Health. 2019;19(1):1247.
2. Maslach C. Job Burnout:New Directions in Research and Intervention. Current Directions in Psychological Science. 2003;12(5):189-192.
3. Shanafelt TD, Hasan O, Dyrbye LN, Sinsky C, Satele D, Sloan J, West CP. Changes in Burnout and Satisfaction With Work-Life Balance in Physicians and the General US Working Population Between 2011 and 2014. Mayo Clin Proc. 2015;90(12):1600-1613.
4. Williams ES, Konrad TR, Scheckler WE, Pathman DE, Linzer M, McMurray JE, Gerrity M, Schwartz M. Understanding Physicians' Intentions to Withdraw from Practice: The Role of Job Satisfaction, Job Stress, Mental and Physical Health. Health Care Management Review. 2001;26(1).
5. Ramirez AJ, Graham J, Richards MA, Cull A, Gregory WM, Leaning MS, Snashall DC, Timothy AR. Burnout and psychiatric disorder among cancer clinicians. British Journal of Cancer. 1995;71(6):1263-1269.
6. Goldberg R, Boss RW, Chan L, Goldberg J, Mallon WK, Moradzadeh D, Goodman EA, McConkie ML. Burnout and Its Correlates in Emergency Physicians: Four Years' Experience with a Wellness Booth. Academic Emergency Medicine. 1996;3(12):1156-1164.
7. Rotenstein LS, Torre M, Ramos MA, Rosales RC, Guille C, Sen S, Mata DA. Prevalence of Burnout Among Physicians: A Systematic Review. Jama. 2018;320(11):1131-1150.
8. Shanafelt TD, Sloan JA, Habermann TM. The well-being of physicians. Am J Med. 2003;114(6):513-519.
9. Hall LH, Johnson J, Watt I, Tsipa A, O'Connor DB. Healthcare Staff Wellbeing, Burnout, and Patient Safety: A Systematic Review. PLoS One. 2016;11(7):e0159015.
10. DiMatteo MR, Sherbourne CD, Hays RD, Ordway L, Kravitz RL, McGlynn EA, Kaplan S, Rogers WH. Physicians' Characteristics Influence Patients' Adherence to Medical Treatment: Results From the Medical Outcomes Study. Health Psychology. 1993;12(2):93-102.
11. Van der Heijden B, Brown Mahoney C, Xu Y. Impact of Job Demands and Resources on Nurses' Burnout and Occupational Turnover Intention Towards an Age-Moderated Mediation Model for the Nursing Profession. Int J Environ Res Public Health. 2019;16(11).
12. Solms L, van Vianen A, Koen J, Theeboom T, de Pagter APJ, De Hoog M, Challenge, Support Research N. Turning the tide: a quasi-experimental study on a coaching intervention to reduce burn-out symptoms and foster personal resources among medical residents and specialists in the Netherlands. BMJ Open. 2021;11(1):e041708.
13. Melnyk BM, Kelly SA, Stephens J, Dhakal K, McGovern C, Tucker S, Hoying J, McRae K, Ault S, Spurlock E, Bird SB. Interventions to Improve Mental Health, Well-Being, Physical Health, and Lifestyle Behaviors in Physicians and Nurses: A Systematic Review. Am J Health Promot. 2020;34(8):929-941.
14. Rock D, Siegel DJ, Poelmans SAY, Payne J. The Healthy Mind Platter. NeuroLeadershipjournal. 2012(4):1-23.
15. Baik SH, Fox RS, Mills SD, Roesch SC, Sadler GR, Klonoff EA, Malcarne VL. Reliability and validity of the Perceived Stress Scale-10 in Hispanic Americans with English or Spanish language preference. J Health Psychol. 2019;24(5):628-639.
16. Lee B, Jeong HI. Construct validity of the perceived stress scale (PSS-10) in a sample of early childhood teacher candidates. Psychiatry and Clinical Psychopharmacology. 2019;29(1):76-82.

ELIGIBILITY:
Inclusion Criteria:

* Employee, student, trainee or volunteer at the Erasmus University Medical Center
* 18-66 years old

Exclusion Criteria:

* Inadequate comprehension of the Dutch language

Ages: 18 Years to 66 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-01-01 (Estimated); Study Completion 2024-01-01 (Estimated)

PRIMARY OUTCOMES:
PSS-10 | T=0 months, T=3 months, T=6 months
  Perceived stress scale 10

SECONDARY OUTCOMES:
Vita-16 | T=0 months, T=3 months, T=6 months
  Vitality scale
Hair cortisol | T=0 months, T=3 months
  Concentration of cortisol in hair. Measurement of longterm stress

OTHER OUTCOMES:
Other study parameters | T=0 months, T=3 months, T=6 months
  Age, gender, profession, department, fulltime/part-time employment, use of corticosteroids, intoxications, hair characteristics, use of Your World among colleagues. After the study period we will also ask participants to evaluate the app. Study parameters collected from the Your World app: use of the Your World app, vitality scores, mood scores, challenges started and completed

CONTACTS AND LOCATIONS:
Locations (1):
- Erasmus MC, University Medical Center Rotterdam, Rotterdam, South Holland, Netherlands

IPD SHARING:
Plan to Share IPD: No
Data available upon reasonable request.